## University of New Mexico Health Sciences Center Informed Consent Cover Letter for Survey

## STUDY TITLE

## Enhancing Cancer Prevention and Control Pathways in the Zuni Pueblo - Native Health Initiative

Dr. Shiraz Mishra from the UNM Cancer Center is conducting a research study to improve health among American Indian adults. You are being asked to participate in this study because you are a Native American person who is the right age for certain cancer screening(s).

Your participation will involve a one-time survey, which should take about 20 minutes to complete. Your involvement in the study is voluntary, and you may choose not to participate. You may also withdraw at any time. Your decision to participate will have no impact upon the care you receive.

The survey includes questions about yourself, your thoughts, feelings and preferences related to healthcare as well as your impression regarding factors that affect delivery of cancer screening services and strategies that can help sustain screening in the community. You can refuse to answer any of the questions at any time. There are no names or identifying information associated with the survey.

There is a very small risk of loss of privacy/confidentiality. Also, some individuals may experience discomfort when answering questions. All data will be kept for 3 years in a locked file in Dr. Mishra's office and in password-protected computer files and then destroyed.

The findings from this project will provide information to improve cancer screening services in the Zuni community. If the research is published, the results will be presented in summary form only, and without your name or any personally identifiable information.

In return of your time, you will receive a \$25 merchandise card completing the survey.

If you have any questions about this research project, please feel free to call Dr. Shiraz Mishra at (505) 925-6085. If you have questions regarding your legal rights as a research participant, you may call the UNMHSC Office of Human Research Protections at (505) 272-1129.

If you complete the survey, you agree to take part in this research study.

Thank you for your consideration.

Sincerely,

Shiraz I. Mishra, MBBS, PhD Professor, UNM Cancer Center and the Department of Pediatrics

HRRC #18-264 Page 1 of 1 Consent: Survey, Version 1, June 15, 2018